CLINICAL TRIAL: NCT01715259
Title: A Phase 1 Single Dose Open-Label Reduced/Staged Pharmacokinetic Study of Abiraterone Acetate in Male Subjects With Impaired Renal Function Compared to Matched Control Subjects With Normal Renal Function
Brief Title: A Pharmacokinetic Study of Abiraterone Acetate in Male Participants With Impaired Renal Function Compared to Individuals With Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cougar Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016951; COU-AA-012 (Other: Cougar Biotechnology, Inc.)
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Renal Insufficiency
Keywords: Renal insufficiency; Renal impairment; End-stage renal disease; Abiraterone acetate; Pharmacokinetics
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abiraterone acetate (Experimental)
  Interventions: Drug: Abiraterone acetate: participants with end-stage renal disease; Drug: Abiraterone acetate: matched control participants with normal renal function

INTERVENTIONS:
Drug: Abiraterone acetate: participants with end-stage renal disease — abiraterone acetate 1000 mg (4 x 250 mg tablets) taken by mouth as a single dose in the fasted state on Day 1
Drug: Abiraterone acetate: matched control participants with normal renal function — abiraterone acetate 1000 mg (4 x 250 mg tablets) taken by mouth as a single dose in the fasted state on Day 1

SUMMARY:
The purpose of this study is to determine the pharmacokinetic (how the drug concentrations change over time) profile of abiraterone acetate 1000 mg when administered as a single dose in male participants with impaired renal function compared to individuals with normal renal function.

DETAILED DESCRIPTION:
This is an open-label (identity of assigned study drug will be known) pharmacokinetics study evaluating a single dose of abiraterone acetate 1000 mg administered in male participants with end-stage renal disease compared to matched-control (matched for age and body mass index) participants with normal renal function. There will be approximately 8 participants in each cohort (group). The total study duration for each participant will be 36 days. Abiraterone acetate 1000 mg will be administered orally (by mouth) as a single dose in the fasted state on Day 1. No food will be ingested for 4 hours post-dose. Participants will be confined to the clinical research center from the day prior to dosing (Day -1) to Day 5 and will return to the clinic on Days 8, 15, and 22 for follow up. Serial pharmacokinetic samples will be collected and safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* Non-smokers or light smokers
* Body Mass Index of 18-38 kg/m2 inclusive
* Negative drug test, at screening and Day -1, for breathalyzer alcohol and drugs of abuse
* Negative HIV antibody test at screening
* Clinical laboratory values within protocol-defined parameters
* Agrees to protocol-defined use of effective contraception
* Participants may have concurrent stable medical conditions and may be included if the deemed condition(s) will not introduce an additional risk factor and will not interfere with the study objectives and procedures

Patients with renal impairment must additionally meet the following criteria:

* Must have protocol-defined criteria of end-stage renal disease, moderate or mild renal impairment
* Evidence of stable renal impairment

Control participants with normal renal function must additionally meet the following criteria:

- Must be in good health

Exclusion Criteria:

All participants:

* Medical history of malignancy except non-melanoma skin cancer
* Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives of that drug or 30 days prior to dosing with abiraterone acetate, whichever is longer
* History of alcoholism or drug abuse within the past 12 months
* Significant history or clinical manifestation as determined by the Investigator of any significant metabolic, allergic, dermatological, hepatic, hematological, pulmonary, cardiovascular, immunologic, neurological, psychiatric or gastrointestinal conditions, surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs
* Clinically significant arrhythmias and/or history or presence of a clinically significantly abnormal electrocardiogram
* Acute illness, especially any active and uncontrolled infection
* Not willing to refrain from strenuous exercise from 48-hours prior to Day -1 and during the period of confinement at the clinical site
* Not willing to abstain from consuming: grapefruit- or caffeine-containing foods or beverages for 72 hours prior to Day -1 and alcohol-containing foods or beverages for 24 hours prior to Day -1
* Donation of blood or significant loss of blood within 56 days prior to Day 1 or planned donation of blood or plasma from screening through 30 days after Day 1, inclusive
* The use of any prescription or over-the-counter (OTC) preparation known to significantly inhibit or induce liver enzymes involved in drug metabolism within 30 days prior to Day 1
* Use of any prescription medications/products or any OTC, non-prescription preparations unrelated to existing allowable stable medical conditions within 5 half-lives of that product or 7 days prior to dosing with abiraterone acetate, whichever is longer
* Any acute or chronic condition that, in the opinion of the Investigator, would limit the individual's ability to complete and/or participate in this clinical study

Patients with renal impairment who meet any of the following criteria will be excluded from the study:

* Acute or exacerbating renal disease, fluctuating or rapidly deteriorating renal function as indicated by widely varying or worsening of signs of renal impairment within 2 weeks of Day 1
* Hypertension (systolic blood pressure [BP] >180 or diastolic BP >100)

Control participants with normal renal function who meet any of the following criteria will be excluded from the study:

* Hypertension (systolic BP >=160 or diastolic BP >=95)
* Any significant laboratory results consistent with renal impairment

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration of abiraterone | Within 0.5 hour prior to dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours post-dose
Time to maximum plasma concentration of abiraterone | Within 0.5 hour prior to dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours post-dose
Area under the concentration-time curve from time 0 to the last measurable plasma concentration of abiraterone | Within 0.5 hour prior to dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours post-dose
Area under the concentration-time curve from time 0 to infinity of abiraterone | Within 0.5 hour prior to dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours post-dose
Terminal phase rate constant of abiraterone | Within 0.5 hour prior to dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours post-dose
Terminal plasma elimination half-life of abiraterone | Within 0.5 hour prior to dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours post-dose
Oral clearance of abiraterone | Within 0.5 hour prior to dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours post-dose
Apparent volume of distribution of abiraterone | Within 0.5 hour prior to dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours post-dose

SECONDARY OUTCOMES:
Number of participants affected by an adverse event | Up to Day 22

CONTACTS AND LOCATIONS:
Overall Officials: Cougar Biotechnology, Inc. Clinical Trial, Study Director — Cougar Biotechnology, Inc.
Locations (1):
- Orlando, Florida, United States

REFERENCES:
- [Derived] Marbury T, Lawitz E, Stonerock R, Gonzalez M, Jiao J, Breeding J, Haqq C, Verboven P, Stieltjes H, Yu M, Molina A, Acharya M, Chien C, Tran N. Single-dose pharmacokinetic studies of abiraterone acetate in men with hepatic or renal impairment. J Clin Pharmacol. 2014 Jul;54(7):732-41. doi: 10.1002/jcph.253. Epub 2014 Jan 17. PMID 24374856